CLINICAL TRIAL: NCT06556147
Title: A Phase 1 Randomized, Placebo- and Active-controlled, Observer-blind Study in Older Adults With Run-in in Young Adults to Evaluate the Safety, Reactogenicity, and Immunogenicity of Four Dose Levels of VXB-241, A Molecular Clamp Stabilized Prefusion F Glycoprotein Subunit Bivalent Vaccine Candidate for the Prevention of Lower Respiratory Tract Disease Caused by Respiratory Syncytial Virus (RSV) And Human Metapneumovirus (HMPV)
Brief Title: A Study of RSV-HMPV Bivalent Vaccine VXB-241 in Older Adults
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vicebio Australia Proprietary Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: VXB241-001
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers
Keywords: Human Metapneumovirus; Respiratory Syncytial Virus; Vaccine
MeSH Terms: interventions — arexvy

STUDY DESIGN:
Intervention Model Description: Stage 1 is a sequential assignment followed by Stage 2 parallel assignment.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (14):
- Stage 1, Day 1, Sequential Cohort 1 (Experimental): Younger and older adult participants will receive VXB-241 60 mcg (low dose) or Placebo, intramuscularly (IM), once on Day 1.
  Interventions: Biological: VXB-241 60 mcg (Low Dose); Other: Placebo
- Stage 1, Day 1, Sequential Cohort 2 (Experimental): Younger and older adult participants will receive VXB-241 120 mcg (medium dose) or Placebo, IM, once on Day 1.
  Interventions: Biological: VXB-241 120 mcg (Medium Dose); Other: Placebo
- Stage 1, Day 1, Sequential Cohort 3 (Experimental): Younger and older adult participants will receive VXB-241 240 mcg (medium-high dose) or Placebo, IM, once on Day 1.
  Interventions: Biological: VXB-241 240 mcg (Medium-high Dose); Other: Placebo
- Stage 1, Day 1, Sequential Cohort 4 (Experimental): Younger and older adult participants will receive VXB-241 480 mcg (high dose) or Placebo, IM, once on Day 1.
  Interventions: Biological: VXB-241 480 mcg (High Dose); Other: Placebo
- Stage 2, Day 1, Concurrent Group 1a (Experimental): Older adult participants will receive VXB-241 60 mcg (low dose), IM, once on Day 1.
  Interventions: Biological: VXB-241 60 mcg (Low Dose)
- Stage 2, Day 1, Concurrent Group 1b (Experimental): Older adult participants will receive VXB-241 120 mcg (medium dose), IM, once on Day 1.
  Interventions: Biological: VXB-241 120 mcg (Medium Dose)
- Stage 2, Day 1, Concurrent Group 1c (Experimental): Older adult participants will receive VXB-241 240 mcg (medium-high dose), IM, once on Day 1.
  Interventions: Biological: VXB-241 240 mcg (Medium-high Dose)
- Stage 2, Day 1, Concurrent Group 1d (Experimental): Older adult participants will receive VXB-241 480 mcg (high dose), IM, once on Day 1.
  Interventions: Biological: VXB-241 480 mcg (High Dose)
- Stage 2, Day 1, Concurrent Group 2a (Active Comparator): Older adult participants will receive Arexvy 120 mcg, IM, once on Day 1.
  Interventions: Biological: Arexvy 120 mcg
- Stage 2, Day 1, Concurrent Group 3a (Placebo Comparator): Older adult participants will receive Placebo, IM, once on Day 1.
  Interventions: Other: Placebo
- Group 1e: VXB-241 Revaccination in VXB-241 Recipients (Experimental): Approximately 50% of the older adult participants who received VXB-241 240 mcg, will receive VXB-241 240 mcg, IM, (based on 1 month post 1st IMP injection results), once on Day 364 in the second year of the study.
  Interventions: Biological: VXB-241 240 mcg
- Group 1f: Placebo Revaccination in VXB-241 Recipients (Placebo Comparator): Approximately 50% of the older adult participants who received VXB-241 (any dose level), will receive Placebo, IM, once on Day 364 in the second year of the study.
  Interventions: Other: Placebo
- Group 2b: Placebo Arexvy Revaccination (Placebo Comparator): All older adult participants who received Arexvy 120 mcg will receive Placebo revaccination, IM, once on Day 364 in the second year of the study.
  Interventions: Other: Placebo
- Group 3b: VXB-241 (Experimental): All older adult participants who received Placebo will receive VXB-241 240 mcg (based on 1 month post 1st IMP injection results), IM, once on Day 364 in the second year of the study.
  Interventions: Biological: VXB-241 240 mcg

INTERVENTIONS:
Biological: VXB-241 60 mcg (Low Dose) — VXB-241 low dose, single, IM injection.
  Arms: Stage 1, Day 1, Sequential Cohort 1; Stage 2, Day 1, Concurrent Group 1a
Biological: VXB-241 120 mcg (Medium Dose) — VXB-241 medium dose, single, IM injection.
  Arms: Stage 1, Day 1, Sequential Cohort 2; Stage 2, Day 1, Concurrent Group 1b
Biological: VXB-241 240 mcg (Medium-high Dose) — VXB-241 medium-high dose, single, IM injection.
  Arms: Stage 1, Day 1, Sequential Cohort 3; Stage 2, Day 1, Concurrent Group 1c
Biological: VXB-241 480 mcg (High Dose) — VXB-241 high dose, single, IM injection.
  Arms: Stage 1, Day 1, Sequential Cohort 4; Stage 2, Day 1, Concurrent Group 1d
Biological: VXB-241 240 mcg — VXB-241 240 mcg (RSV preF 120 mcg + hMPV preF 120 mcg) (based on 1 month post 1st IMP injection results) single, IM injection.
  Arms: Group 1e: VXB-241 Revaccination in VXB-241 Recipients; Group 3b: VXB-241
Other: Placebo — Placebo, single, IM injection.
  Arms: Group 1f: Placebo Revaccination in VXB-241 Recipients; Group 2b: Placebo Arexvy Revaccination; Stage 1, Day 1, Sequential Cohort 1; Stage 1, Day 1, Sequential Cohort 2; Stage 1, Day 1, Sequential Cohort 3; Stage 1, Day 1, Sequential Cohort 4; Stage 2, Day 1, Concurrent Group 3a
Biological: Arexvy 120 mcg — Arexvy 120 mcg, single, IM injection.
  Arms: Stage 2, Day 1, Concurrent Group 2a

SUMMARY:
The main purposes of this study are to assess the safety, reactogenicity and immunogenicity of 4 dose levels of the bivalent combination Respiratory Syncytial Virus (RSV) / human Metapneumovirus (hMPV) vaccine candidate VXB-241 when administered as a single-dose regimen to healthy adults 60 to 83 years of age, and to assess the impact of revaccination approximately 1 year later.

DETAILED DESCRIPTION:
This is a multi-center study in older adults with run-in in younger adults to evaluate the safety, reactogenicity, and immunogenicity of 4 dose levels of VXB-241. The total planned sample size is 136 randomized participants, composed of 16 younger adults 18 to 40 years of age and 120 older adults 60 to 83 years of age who are in good health, which allows for many chronic conditions, if well controlled and compatible with self-sufficiency in self-care and daily living activities.

Recruitment will be in 2 stages:

* Stage 1 (Sequential Cohort Stage, N=32). Four cohorts (Cohorts 1 to 4), each of 8 participants, will be enrolled sequentially. In each cohort, 4 younger adults will be enrolled first, followed by 4 older adults. Younger and older adult participants will be randomized with 3:1 ratio to VXB-241 at increasing dose (60 microgram (mcg), 120 mcg, 240 mcg, 480 mcg in Cohorts 1 to 4, respectively) or Placebo. A Safety Monitoring Committee will make recommendations on escalation from one cohort to the next and from Stage 1 to Stage 2 based on safety and reactogenicity data collected over 1 week after investigational medicinal product (IMP) dosing.
* Stage 2 (Concurrent Group Stage, N=104). Older adult participants will be randomized concurrently with unequal randomization to 1 of 6 treatment groups: VXB-241 60 mcg (Group 1a), VXB-241 120 mcg (1b), VXB-241 240 mcg (1c), VXB-241 480 mcg (1d), commercial RSV vaccine Arexvy (2a), Placebo (3a). The planned total sample size of each treatment group, combining Stage 1 and Stage 2, is N=20.

The overall planned duration of the study is approximately 6 months for younger adult participants and approximately 2 years for older adult participants.

At the end of the 1st year, older adult participants will receive a second IMP injection (revaccination): participants who received VXB-241 (at any dose) will be assigned 1:1 to revaccination with VXB-241 (Group 1e) or Placebo (1f); participants who received Arexvy will be revaccinated with placebo (2b); participants who received Placebo will be revaccinated with VXB-241 (3b). The dose of VXB-241 for revaccination will be 240 mcg (RSV preF 120 mcg + HMPV preF 120 mcg) (based on 1 month post 1st IMP injection results).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 40 years of age (yoa) (younger adult) or 60 to 83 yoa (older adult).
2. Evidence of signed and dated participant informed consent form (PICF) prior to any study procedure, indicating that the participant has been informed of all pertinent aspects of the study.
3. Willingness and ability to comply with the planned study visits and calls, procedures, and restrictions for the duration of the study.
4. Good health, which allows for pre-existing well-controlled and low impact chronic diseases, except for the diseases listed in the exclusion criteria. A disease is defined as well-controlled and low impact if it did not require meaningful change in therapy or unplanned medical visits in the previous 3 months and allows participant's primary responsibility for self-care and daily living activities.
5. Non-smoker or occasional smoker, defined as smoking less than 10 nicotine-containing cigarettes/ vapes/cigars/pipe fills per week.
6. Contraception: heterosexually active participants of childbearing potential able and willing to use a double contraceptive method for at least 4 weeks before and 12 weeks after the first IMP injection at Visit 2 (all participants of childbearing potential) and second IMP injection at Visit 6 (male older adults of childbearing potential).
7. Body Mass Index (BMI) >=17.0 kilogram per square meter (kg/m^2) and less than or equal to (<=) 35.0 kg/m^2.

Exclusion Criteria:

1. History of RSV and/or hMPV infection affecting the participant and/or the participant's household in the previous 12 months.
2. History of autoimmune disease (AID) or potentially autoimmune disease (pAID) requiring therapeutic intervention, even if stable and well controlled, including but not limited to systemic lupus erythematosus, autoimmune arthritis/rheumatoid arthritis, Guillain-Barré syndrome, multiple sclerosis, Sjögren's syndrome, idiopathic thrombocytopenia purpura, glomerulonephritis, autoimmune thyroiditis, temporal arteritis, psoriasis, insulin-dependent diabetes mellitus, celiac disease.
3. Confirmed or suspected immunodeficiency, even if stable and well controlled.
4. Ongoing severe asthma. Other allergic diseases (example, allergic rhinitis, atopic dermatitis / eczema, mild to moderate asthma, food allergies, are allowed at the investigator's or delegate's discretion).
5. History of severe allergic reaction (example, anaphylaxis) to any substance, including vaccine components and latex.
6. History of severe adverse event (AEs) associated with vaccine administration.
7. Ongoing disorders of coagulation, which contraindicate IM injections.
8. Donation or loss of >=500 milliliter (mL) whole blood on the previous 2 months and/or donation of plasma in the previous 1 week, and/or intention to donate blood or plasma during the study.
9. Positive serum test results for serum human immunodeficiency virus (HIV), hepatitis B virus (HBV) and/or hepatitis C virus (HCV) infection and/or documented HIV, HVB or HVC infection.
10. Other poorly controlled and/or impactful chronic disease. A disease is defined as poorly controlled if it required meaningful change in therapy and/or unplanned medical visits in the previous 3 months. A disease is defined as impactful if it has a meaningful impact on participant's self-care and/or activities of daily living.
11. Disease expected to prevent completion of the study (that is to rapidly deteriorate within the timeframe of the study).
12. Prior treatments.

    1. Licensed RSV vaccine or investigational RSV and/or hMPV vaccine received at any time.
    2. Investigational drug or vaccine received in the previous 6 months.
    3. Chemotherapy, radiotherapy, and/or other immunosuppressive medication including biologics received in the previous 6 months.
    4. Immunoglobulins G (IgGs) or any blood product received in the previous 3 months.
    5. Systemic corticosteroids (oral/intravenous/intramuscular) at doses equivalent to >=20 mg prednisone received for >=14 days, even if not consecutive, during the previous 3 months. Inhaled/nebulized, intra-articular, intra-bursal, skin and eye topical corticosteroids are permitted.
13. Clinically meaningful abnormal finding from physical examination, vital sign assessment, electrocardiogram (ECG), safety laboratory test results. If deemed appropriate, the investigator or delegate may repeat these assessments.
14. History of alcohol abuse in the previous year and/or positive alcohol breath test.
15. History of recreational drug abuse in the previous year and/or positive test for drugs of abuse, unless there is an explanation acceptable to the investigator (example, the participant has informed in advance that he/she consumed a prescription or over-the-counter product that contained the detected drug).
16. Intention to participate in any investigational drug/vaccine clinical trial at any time throughout the planned duration of this study.
17. Presence of tattoo, scarring, skin discoloration, or any other skin disturbances at the injection site which may interfere with effective assessment of the injection site.
18. Intention to move to a location that would prevent participating in the study until study end.
19. Limited to premenopausal female participants: breastfeeding, positive pregnancy test or intention to become pregnant during the first 3 months of the study.
20. Any other reason which would prevent the participant from participating in the study or interfere with the participant's compliance with study procedures.

Ages: 18 Years to 83 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2024-08-13 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of Older Adult Participants With 1 or More Unsolicited AEs | 1 month after first IMP injection (Days 1 to 30)
Proportion of Older Adult Participants With 1 or More Solicited AEs | 7 days after first IMP injection (Days 1 to 8)
Geometric Mean Fold Increase (GMFI) of RSV-A, RSV-B, hMPV-A, and hMPV-B Serum Neutralizing Antibody Titers in Older Adults | Pre-injection baseline to 1 month (Day 30) after first IMP injection
  GMFI is defined as geometric mean of ratios of specific antibody titer/concentration at each post-vaccination time point over pre-vaccination baseline.
Ratio of Dose-response Curves for GMFIs of RSV-A, RSV-B, hMPV-A and hMPV-B Serum Neutralizing Antibody Titers in Older Adults | Pre-injection baseline to 1 month (Day 30) after first IMP injection
  Ratio of VXB-241 dose versus GMFI of RSV-A, RSV-B, hMPV-A and hMPV-B will be calculated.

SECONDARY OUTCOMES:
Proportion of Older Adult Participants With 1 or More Unsolicited AEs and With 1 or More Severe Unsolicited AE | 1 month after first IMP injection (Days 1 to 30) and 1 month after second IMP injection (revaccination, Days 364 to 394)
Proportion of Older Adult Participants With Serious Adverse Events (SAEs), AEs of Special Interest (AESIs), and Premature Discontinuation Associated AEs (PDAEs) | 1 month after first IMP injection (Days 1 to 30) and 1 month after second IMP injection (revaccination, Days 364 to394), and throughout follow-up (Days 1 to 720)
Mean Change From Baseline for Abnormal and Severe Abnormal Hematology Laboratory Values for Hemoglobin in Older Adults | 7 days (Day 8) and 1 month (Day 30) after first IMP injection, and 1 month (Day 394) after second IMP injection (revaccination
Mean Change From Baseline for Abnormal and Severe Abnormal Hematology Laboratory Values for Red Blood Cells, White Blood Cells, and Platelet Count in Older Adults | 7 days (Day 8) and 1 month (Day 30) after first IMP injection, and 1 month (Day 394) after second IMP injection (revaccination
Mean Change From Baseline for Abnormal and Severe Abnormal Blood Chemistry Laboratory Values for Alanine Transaminase (ALT), Aspartate Transaminase (AST), and Alkaline Phosphatase in Older Adults | 7 days (Day 8) and 1 month (Day 30) after first IMP injection, and 1 month (Day 394) after second IMP injection (revaccination
Mean Change From Baseline for Abnormal and Severe Abnormal Blood Chemistry Laboratory Values for Total Bilirubin, Creatinine, and Urea in Older Adults | 7 days (Day 8) and 1 month (Day 30) after first IMP injection, and 1 month (Day 394) after second IMP injection (revaccination
Proportion of Older Adult With Abnormal and Severe Abnormal Values for Hematology Laboratory Parameter | 7 days (Day 8) and 1 month (Day 30) after first IMP injection, and 1 month (Day 394) after second IMP injection (revaccination)
Proportion of Older Adult With Abnormal Values and Severe Abnormal Values for Blood Chemistry Laboratory Parameter | 7 days (Day 8) and 1 month (Day 30) after first IMP injection, and 1 month (Day 394) after second IMP injection (revaccination)
Proportion of Older Adult Participants With Solicited AEs | 7 days after 2nd IMP injection (revaccination, Day 364 to 371)
GMFI of RSV-A, RSV-B, hMPV-A, and hMPV-B Serum Neutralizing Antibody Titers in Older Adults | Pre-injection baseline to 6 months (Day 182) and 12 months (Day 364) after first IMP injection, and 1 month (Day 394), 6 months (Day 546), and 12 months (Day 720) after second IMP injection (revaccination)
Geometric Mean Titers (GMTs) of RSV-A, RSV-B, hMPV-A, and hMPV-B Serum Neutralizing Antibody Titers in Older Adults | Pre-injection baseline to 1 month (Day 30), 6 months (Day 182) and 12 months (Day 364) after first IMP injection, and 1 month (Day 394), 6 months (Day 546), and 12 months (Day 720) after second IMP injection (revaccination)
Proportion of Older Adult Participants with Sero-response Greater Than or Equal to (>=) 4-fold (SRR-4) and 8-fold (SRR-8) Increase from Baseline in Neutralizing Antibody Titers for RSV-A, RSV-B, hMPV-A and hMPV-B | Pre-injection baseline up to 1 month (Day 30), 6 months (Day 182) and 12 months (Day 364) after first IMP injection, and 1 month (Day 394), 6 months (Day 546), and 12 months (Day 720) after second IMP injection (revaccination)
GMFI of RSV Pre-fusion Protein (Pre-F) and hMPV Pre-F Serum Immunoglobulins G (IgG) Concentrations in Older Adults | Pre-injection baseline up to 1 month (Day 30), 6 months (Day 182) and 12 months (Day 364) after first IMP injection, and 1 month (Day 394), 6 months (Day 546), and 12 months (Day 720) after second IMP injection (revaccination)
Geometric Mean Concentrations (GMC) of Serum IgG Versus RSV Pre-F and hMPV Pre-F in Older Adults | Up to 1 month (Day 30), 6 months (Day 182), and 12 months (Day 364) after first IMP injection and 1 month (Day 394), 6 months (Day 546) and 12 months (Day 720) after second IMP injection (revaccination)
Geometric Mean Ratios (GMRs) of Fold Increase of RSV-A and RSV-B Neutralizing Serum Antibody Titers Versus Fold Increase of RSV Pre-F Serum IgG Concentration in Older Adults | Pre-injection baseline up to 1 month (Day 30), 6 months (Day 182) and 12 months (Day 364) after first IMP injection, and 1 month (Day 394), 6 months (Day 546), and 12 months (Day 720) after second IMP injection (revaccination)
GMR of Fold Increase of hMPV-A and hMPV-B Neutralizing Serum Antibody Titers Versus Fold Increase of hMPV Pre-F Serum IgG Concentration in Older Adults | Pre-injection baseline up to 1 month (Day 30), 6 months (Day 182) and 12 months (Day 364) after first IMP injection, and 1 month (Day 394), 6 months (Day 546), and 12 months (Day 720) after second IMP injection (revaccination)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nischal Sahai, Principal Investigator — University of the Sunshine Coast; Dr. Stephanie Wallace, Principal Investigator — University of the Sunshine Coast; Dr. Christopher Moller, Principal Investigator — University of the Sunshine Coast; Dr. Ian Forsyth, Principal Investigator — Veritus Research
Locations (4):
- Australia (4):
  - University of the Sunshine Coast, Morayfield, Queensland
  - University of the Sunshine Coast, Sippy Downs, Queensland
  - University of the Sunshine Coast, South Brisbane, Queensland
  - Veritus Research, Bayswater, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Young A, Kolekar S, Mendoza CA, Jaberolansar N, Modhiran N, Webb T, McCuaig R, Kommajosyula V, Tardiota N, Dy Q, Amarilla AA, Dalrymple RL, Gillard M, Dutton JL, Magdalena J, Vandendriessche F, Smal J, Young PR, Watterson D, Hanon EJ, Chappell KJ. A second-generation molecular clamp stabilised bivalent candidate vaccine for protection against diseases caused by respiratory syncytial virus and human metapneumovirus. PLoS Pathog. 2025 Jul 17;21(7):e1013312. doi: 10.1371/journal.ppat.1013312. eCollection 2025 Jul. PMID 40674411